CLINICAL TRIAL: NCT03456310
Title: Role of Transperineal Ultrasonography on Basis of Dynamic Pelvic MRI in Diagnosis of Female Pelvic Floor Dysfunction.
Brief Title: Transperineal US on Basis of MRI in Female Pelvic Floor Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AShassan, Assistant lecturer-radiology department-assiutU, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TPUS MRI PELVIC FLOOR
Record Dates: First submitted 2018-02-21; First posted 2018-03-07 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trans-perineal ultrasound (Experimental): Transperineal ultrasonography is done by 2D ultrasound machine, curved probe is placed in the perineum, mid sagittal and axial views are obtained Then it's accuracy is assessed according to findings on dynamic pelvic MRI .
  Interventions: Diagnostic Test: transperineal ultrasound

INTERVENTIONS:
Diagnostic Test: transperineal ultrasound — trans-perineal US: B mode capable 2D ultrasound system with cine loop function, a 3.5-6.0 MHz curved array transducer. A mid-sagittal and axial views is obtained by placing a transducer on the perineum (Parting of the labia can improve image quality).
  Dynamic MRI:
  Magnetic resonance (MR) imaging of the pelvic floor is a two-step process that includes:
  analysis of anatomic damage on axial fast spin-echo (FSE) T2-weighted images. then sagittal and coronal (FSE) T2-weighted are obtained.
  functional evaluation using sagittal dynamic single-shot T2-weighted sequences during straining and defecation.
  Other Names: dynamic pelvic MRI

SUMMARY:
Pelvic floor failure is a common disorder that can seriously jeopardize a woman's quality of life by causing urinary and fecal incontinence, difficult defecation and pelvic pain. Multiple congenital and acquired risk factors are associated with pelvic floor failure, including altered collagen metabolism, female sex, vaginal delivery, menopause and advanced age. A complex variety of fascial and muscular lesions that range from stretching, insertion detachment, denervation atrophy and combinations of pelvic floor relaxation to pelvic organ prolapse may manifest in a single patient.

The prevalence of pelvic floor dysfunction increases with age. It is approximately 9.7% in child bearing period (20-39 yrs), while it reaches up to 49.7% by 80 yrs and older. Thorough preoperative assessment of pelvic floor failure is necessary to reduce the rate of relapse, which is reported to be as high as 30%.

MR imaging is a powerful tool that enables radiologists to comprehensively evaluate pelvic anatomic and functional abnormalities, thus helping surgeons provide appropriate treatment and avoid repeat operations.

Real time 2D trans-perineal ultrasound is emerging as an exciting new technique for pelvic floor assessment. It has advantage of providing a global view of the entire pelvic floor, from the symphysis to the ano-rectum, and includes the lower aspects of the levator ani muscle, in addition to its lower costs and greater accessibility; also sonographic imaging is more useful in the clinical environment, and generally better tolerated than magnetic resonance imaging.

DETAILED DESCRIPTION:
Patient: 135 female patients in child bearing period (20-39 yrs) will undergo trans-perineal ultrasound and dynamic pelvic MRI:

40 days after vaginal delivery or cesarean section for asymptomatic and symptomatic cases.

revision after six months for cases with sonongraphic or MRI findings. after obtaining an informed written consent and approval of the ethical committee of faculty of medicine of Assiut University.

Inclusion criteria: asymptomatic and symptomatic female Patients in child bearing period 40 days after vaginal delivery and cesarean section.

Exclusion criteria: patients with previous pelvic floor surgery.

Patient preparation

For trans-perineal US:

- Patient is positioned in dorsal lithotomy position, with the hips flexed and slightly abducted and after bladder and bowel emptying. The pelvic tilt can be improved by asking the patient to place their heels as close as possible to the buttocks and move hips towards the heels.

For MRI:

- Patient is positioned in supine position and using pelvic coil after bladder and bowel emptying.

Method:

1. trans-perineal US: B mode capable 2D ultrasound system with cine loop function, a 3.5-6.0 MHz curved array transducer. At women health hospital. A mid-sagittal and axial views is obtained by placing a transducer on the perineum (Parting of the labia can improve image quality).

   The following measures will be obtained:

   Hiatus diameter, bladder neck descent, and descent of other pelvic organs in relation to reference line (parallel to lower part of public bone).
2. Dynamic MRI:

Magnetic resonance (MR) imaging of the pelvic floor is a two-step process that includes:

analysis of anatomic damage on axial fast spin-echo (FSE) T2-weighted images. then sagittal and coronal (FSE) T2-weighted are obtained.

functional evaluation using sagittal dynamic single-shot T2-weighted sequences during straining and defecation to show descent of pelvic organs and pelvic floor relaxation or weakness.

ELIGIBILITY:
Inclusion Criteria:

* asmptomatic and symptomatic female Patients in child bearing period 40 days after vaginal delivery and cesarean section.

Exclusion Criteria:

* patients with previous pelvic floor surgery.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 135 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
role of trans-perineal ultrasound in diagnosis of pelvic floor dysfunction | 4 years
  accuracy of trans-perineal ultrasound in detection and assessment of female pelvic floor dysfunction